CLINICAL TRIAL: NCT00145184
Title: Effect of Multivitamin Supplements on Clinical and Immunological Response in Childhood Tuberculosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-117; NCT00197535 (obsolete NCT alias)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Tuberculosis
Keywords: multivitamin, supplements, tuberculosis, Tanzania
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Multivitamins (Experimental): Multivitamin supplement containing the following vitamins: B1, B2, Niacin, B6, Folate, B12, C, and E
  Interventions: Dietary Supplement: Multivitamin supplement containing vitamins B, C, and E

INTERVENTIONS:
Dietary Supplement: Multivitamin supplement containing vitamins B, C, and E — A daily oral dose of between 1.5 to 3 times the age- appropriate Recommended Dietary Allowance (RDA) of each vitamin taken for two months starting at enrollment.
  Arms: Multivitamins
Drug: Placebo — Placebo pill taken orally once per day for two months starting at enrollment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see whether children who take vitamins along with the standard medicine for tuberculosis (TB) recover better and quicker than children who take only the standard medicine for TB. Four hundred children ages 6 weeks-5 years, who have been diagnosed with tuberculosis, will be enrolled. They will be followed for 2 months after treatment for TB. Study procedures may include blood draws, Tuberculin Skin Tests, body measurements, gastric aspirates (removal of stomach fluid), physical exams, and questionnaires. This study will occur in Tanzania.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the single most common infectious disease cause of mortality worldwide with evidence that support nutritional status may be associated with poor outcomes in TB patients. Data from observational and limited intervention studies support the hypothesis that nutritional supplements/micronutrients may be beneficial as well as potential treatments in TB. The effect of micronutrient status will be examined in the context of a double blinded placebo controlled randomized trial; 400 tuberculosis patients (age 6 weeks to 5 years) will be randomized to receive either multi-micronutrients or placebo from the start of their anti-TB therapy, through 2 months of their anti-TB therapy. The primary objective is to evaluate the efficacy of a multivitamin supplement containing vitamins B, C and E on weight gain in childhood tuberculosis at 2 months after start of anti-tuberculosis therapy. Secondary objectives are to: evaluate the efficacy of a multivitamin supplement containing vitamins B, C, and E on clearance of chest x-ray in childhood tuberculosis at 2 months after start of anti-tuberculosis therapy; compare the treatment arms with respect to the following immunological parameters: ex-vivo lymphocyte proliferation; cytokines production including IL-2, IL-12, TNF - alpha, INF-gamma; and CD4 and CD8 T-lymphocyte counts at 2 months after start of anti-tuberculosis therapy; assess the validity of Tuberculin Skin Test (TST) for the diagnosis of childhood tuberculosis in a population with high BCG coverage and HIV prevalence; assess the validity and feasibility of using "microscopic observation broth drug susceptibility (MODS) assay" of sputum and gastric aspirates in the diagnosis of childhood tuberculosis; correlate the above-mentioned immunological markers (IL-2, IL-12, INF-gamma and TNF-alpha) with weight gain and chest x-ray at 2 months after start of anti-tuberculosis therapy; and compare the immunological response to a supplement containing vitamins B, C and E in childhood tuberculosis patients with and without HIV infection. The endpoints of interest include immunological parameters like CD4 T lymphocyte count and clinical outcomes such as, weight gain and resolution of chest x-ray after 2 months anti-TB therapy. Researchers will also examine the utility of these immune response parameters as surrogate markers for treatment efficacy in TB, irrespective of nutritional and other risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Loss of more than 10% of maximum weight or failure to gain weight for 2 months.
* Having cough with wheeze for 4 weeks or more.
* History of household contact with a probable or confirmed tuberculosis case in the past 6 months.
* Pyrexia of unknown origin.
* Painless swelling in a group of cervical lymph nodes.
* Children who were diagnosed with TB in the past 5 years and have received anti-tuberculosis therapy for a period less than 4 weeks.

Exclusion Criteria:

-Children who have been treated with anti-tuberculosis therapy exceeding 4 weeks in the past one year will not be eligible for entry into the study

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
weight gain in childhood tuberculosis | 2 months after start of anti-tuberculosis therapy.

SECONDARY OUTCOMES:
clearance of chest x-ray in childhood tuberculosis | 2 months after start of anti-tuberculosis therapy
immunological parameters: ex-vivo lymphocyte proliferation; cytokines production including IL-2, IL-12, TNF - alpha, interferon-gamma; and CD4 and CD8 T-lymphocyte counts | 2 months after start of anti-tuberculosis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimbili University, College of Health Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Mehta S, Mugusi FM, Bosch RJ, Aboud S, Chatterjee A, Finkelstein JL, Fataki M, Kisenge R, Fawzi WW. A randomized trial of multivitamin supplementation in children with tuberculosis in Tanzania. Nutr J. 2011 Oct 31;10:120. doi: 10.1186/1475-2891-10-120. PMID 22039966